CLINICAL TRIAL: NCT03913884
Title: Effect of Concentrated Growth Factor (CGF) on Short Term Clinical Outcomes After Partially Impacted Mandibular Third Molar Surgery: A Split-Mouth Randomized Clinical Study
Brief Title: Effect of CGF on Short Term Clinical Outcomes After Partially Impacted Mandibular Third Molar Surgery
Acronym: CGF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Işık, Oral Surgery, Ege University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: Faculty of Dentistry
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain; Trismus; Edema
Keywords: Impacted third molar surgery; Clinical outcomes; Concentrated growth factor
MeSH Terms: conditions — Pain, Postoperative; Trismus; Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentrated growth factor Group (Experimental): Group I (test); in which CGF fibrin matrix was applied to the extraction socket
  Interventions: Procedure: Concentrated growth factor
- Non-Concentrated growth factor Group (Experimental): Group II (control); in which CGF was not applied to the extraction socket
  Interventions: Other: Non-Concentrated growth factor Group

INTERVENTIONS:
Procedure: Concentrated growth factor — CGF fibrin matrix was placed in one socket which was randomly selected (test side). The flap was sutured with 4/0 atraumatic silk suture (½ cutting edge, 75 cm, Doğsan, İstanbul, Turkey) for each surgical site.
  Arms: Concentrated growth factor Group
Other: Non-Concentrated growth factor Group — To control group, extraction of the tooth on the opposite site was performed and the socket left to heal naturally. The flap was sutured with 4/0 atraumatic silk suture (½ cutting edge, 75 cm, Doğsan, İstanbul, Turkey) for each surgical site.
  Arms: Non-Concentrated growth factor Group

SUMMARY:
The aim of this study was to evaluate the effectiveness of concentrated growth factor (CGF) on soft tissue healing and postoperative side effects following third molar surgery. This study was designed on 60 patients as a randomized single-blind clinical trial. The predictor variable was the implementation of CGF fibrin matrix, which was categorized as CGF and non-CGF. The primary outcome variable of the study was the healing of soft tissue around the extraction socket. The secondary outcome variables were pain, swelling and trismus. Data were analyzed using the non-parametric Brunner and Langer model. Statistical significance was set at P < .001.

DETAILED DESCRIPTION:
The study population was composed of subjects presenting to the Department of Oral Surgery for evaluation and management of bilateral, partially-impacted mandibular third molars. The protocol for this study was approved by the local ethics committee and all participants signed an informed consent.

A patient who was referred for extraction of mandibular third molars was examined clinically and radiologically according to the inclusion criteria.

Before the partially-impacted mandibular third molar surgery, randomisation was achieved by use of sealed envelopes, selected by the patient. The envelopes contained cards labelled 'right' or 'left', which indicated the surgical side to receive CGF application.The envelopes were opened by the surgeon after the patients made their selection.

Both partially-impacted mandibular third molars were extracted by the same experienced surgeon. For each patient, the sites operated on were randomly divided into two study groups.

Group I (test); in which CGF fibrin matrix was applied to the extraction socket Group II (control); in which CGF was not applied to the extraction socket Each patient was listed for two surgical appointments. The second extraction was done on the control side, three weeks after the first extraction.

Patients were blind as to which side the CGF was placed, in order to avoid any influence on visual analog scale (VAS) scores. To obtain an objective assessment of pain, patients were informed that CGF application was used on all sites by the surgeon. The surgeon was not blind to the CGF application or the suturing. Therefore, clinical parameters were assessed based on the classifications by an independent observer specializing in oral surgery.

Study variables The primary variable of this clinical study was CGF application. CGF Preparation CGF was prepared according to Sacco protocol. The patients' blood was collected in 9 ml glass two tubes with vacutainer. The tubes were centrifuged immediately in a special centrifuge device (Medifuge, France). After the following settings were used: 2 min 2700 rpm, 4 min 2400 rpm, 4 min 2700 rpm and 3 min 3000 rpm, three layers were observed in the tubes. The upper layer, comprising platelet-poor plasma and the lower one, the red blood cells, were separated from the 'buffy coat', the CGF, by forceps and scissors.

The primary outcome variable was soft tissue healing around the extraction socket. The secondary outcome variables were pain, swelling and trismus.

Before surgery, patients rinsed their mouths with 0.12% clorhexidine gluconate as an antiseptic mouthwash for 60 seconds.

All surgeries were carried out using the same protocol by the same experienced surgeon. As local anesthetic, 2% lidocaine with 1:80.000 epinephrine (1/200.000 Jetokain®, Adeka, İstanbul, Turkey) was applied. A mucoperiosteal flap was elevated to expand initial access without releasing. The surgical approach for each tooth was as follows: bone removal, simple mobilization, extraction of tooth without sectioning and curettage of the socket. After extraction, the socket was irrigated using 60 mL of sterile saline.

CGF fibrin matrix was placed in one socket which was randomly selected (test side). After three weeks, extraction of the tooth on the opposite site was performed and the socket left to heal naturally (control side). The flap was sutured with 4/0 atraumatic silk suture (½ cutting edge, 75 cm, Doğsan, İstanbul, Turkey) for each surgical site.

Postoperatively, amoxicillin (500 mg/8 h, Largopen®, Bilim Pharmaceuticals, İstanbul, Turkey for five days), 0.2% chlorhexidine mouthwash (twice per day for seven days; Kloroben®, Drogsan Pharmaceuticals, Ankara, Turkey) and paracetamol (500 mg, every 4-6 h, Parol®, Atabay Pharmaceuticals, İstanbul, Turkey) were prescribed by the surgeon. After one week, sutures were removed.

All subjects were recalled postoperatively at the 3rd and 7th days by the blinded examiner. Soft tissue healing, pain, swelling and trismus were evaluated on the 3rd and 7th days and pain scores, noted from 1st to 7th days by the patient, were collected. Demographic values for patients' age and gender were also noted.

ELIGIBILITY:
Inclusion Criteria:

1- Bilateral, vertically, partially-impacted Class I, Level B third molars

Exclusion Criteria:

1. Infection of the surgical region
2. Smoking habit
3. Alcohol usage
4. Physical or mental disability
5. Thrombocytopenia
6. Chemotherapy in head and neck region
7. Pregnant woman or woman in menstrual cycle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2018-08-26 (Actual)

PRIMARY OUTCOMES:
soft tissue healing | Change of soft tissue healing at 7 days
  This was assessed on the third and seventh preoperative days using the healing index classified by Landry et al.12. It depends on tissue colour, presence of bleeding on palpation, epithelization of wound margins, granulation tissue and suppuration, and rates the degree of healing attained from 'very poor' to 'excellent'.

SECONDARY OUTCOMES:
severity of postoperative pain | Change of postoperative pain at 7 days
  The patients were instructed to note their level of postoperative discomfort and/or pain on the scale, which ranged from 0, indicating no pain, to 100 indicating the worst ever experienced. Paracetamol (500-mg tablets) was prescribed to be taken postoperatively as needed. The patients were asked to fill in the questionnaire as required on a daily basis for 7 days.
presence of swelling | Change of swelling at 7 days
  three facial measurements were taken with milimetric elastic ruler, preoperatively, as described by Kumar et al., on the third and seventh days after extraction. These dimensions were as follows: the from the tragus to the pogonion (TP); from the tragus to the corner of the mouth (TC); and from the lateral corner of the eye to the angle of the mandible (EA).
presence of trismus | Change of trismus at 7 days
  Inter-incisal distance was measured, as a guide point, with a millimeter ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Işık, Principal Investigator — Oral Surgery
Locations (1):
- Ege University, Faculty of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozveri Koyuncu B, Isik G, Ozden Yuce M, Gunbay S, Gunbay T. Effect of concentrated growth factor (CGF) on short-term clinical outcomes after partially impacted mandibular third molar surgery: A split-mouth randomized clinical study. J Stomatol Oral Maxillofac Surg. 2020 Apr;121(2):118-123. doi: 10.1016/j.jormas.2019.07.002. Epub 2019 Jul 9. PMID 31299343